CLINICAL TRIAL: NCT00606060
Title: Safety and Efficacy of Continuous Infusion of Recombinant Factor VIII - Sucrose-formulated (BAY 14 2222) Concentrate in Patients With Hemophilia A Undergoing Major Elective Surgery.
Brief Title: BAY14-2222 Continuous Infusion in Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11486
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Hemophilia
Keywords: Hemophilia,; Continuous Infusion
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Kogenate (BAY14-2222)

INTERVENTIONS:
Drug: Kogenate (BAY14-2222) — 100 IU/mL (250 IU/vial nominal potency) continuous infusion over 6-11 days in 12 patients. 400 IU/mL (1000 IU/vial nominal potency) continuous infusion over 6-11days in 3 patients.

SUMMARY:
Phase III study, to evaluate the efficacy and safety of continuous infusion of rFVIII-FS in the treatment of patients with hemophilia A undergoing major elective surgery by achieving the required therapeutic concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (FVIII:C </=1%)
* No history of FVIII inhibitor formation and no current evidence of inhibitor antibody (Bethesda Assay < 0.6 BU)
* Elective major surgery requiring at least 6 days of rFVIII-FS therapy
* Subjects should have been previously treated with FVIII concentrates for at least 150 exposure days. Previous treatment could have been with any type of rFVIII or with plasma-derived FVIII concentrate or cryoprecipitate

Exclusion Criteria:

* Abnormal renal function (serum creatinine >1.3 mg/dL)
* Any treatments, which may change the clearance of FVIII (dialysis, plasma exchange)
* Anemia (hemoglobin <11 g/dL)
* Known AIDS (HIV seropositive patients may be enrolled)
* Active liver disease (transaminases > 5 times the upper limit of normal)
* History of severe reaction to FVIII concentrates
* Interferon treatment within the last 3 months
* Thrombocytopenia (< 100,000 platelets/mm3) or other known hematological/bleeding problems other than hemophilia A
* Intake of other investigational drugs within 1 month prior to study entry
* Need for pre-medication for FVIII infusions (e.g. antihistamines)
* Diastolic blood pressure >100 mm/Hg, which could not be controlled with antihypertensive medications

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
efficacy of continuous infusion of recombinant Factor VIII - sucrose-formulated (rFVIII-FS) in the treatment of patients with hemophilia A | 28 days

SECONDARY OUTCOMES:
Evaluate the safety of rFVIII-FS. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Tel Litwinsky, Israel